CLINICAL TRIAL: NCT07035041
Title: A Phase 2 Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of D-2570 as Induction Therapy in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Phase 2 Study of D-2570 in Subjects With Moderately to Severely Active Ulcerative Colitis
Acronym: D2570-202
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2570-202
Record Dates: First submitted 2025-05-19; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: UC - Ulcerative Colitis; Moderately to Severely Active Ulcerative Colitis
Keywords: Moderately to Severely Active Ulcerative Colitis; UC
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- D-2570 (experimental arm 1) (Experimental): Subjects will then be randomized in a 1:1:1 ratio to D-2570 (experimental arm 1), D-2570 (experimental arm 2), or placebo (control arm). They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.
  Interventions: Drug: D-2570
- D-2570 (experimental arm 2) (Experimental): Subjects will then be randomized in a 1:1:1 ratio to D-2570 (experimental arm 1), D-2570 (experimental arm 2), or placebo (control arm). They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.
  Interventions: Drug: D-2570
- placebo (Placebo Comparator): Subjects will then be randomized in a 1:1:1 ratio to D-2570 (experimental arm 1), D-2570 (experimental arm 2), or placebo (control arm). They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-2570 — Subjects will then be randomized in a 1:1:1 ratio to D-2570 or placebo . They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.
  Arms: D-2570 (experimental arm 1); D-2570 (experimental arm 2)
Drug: Placebo — Subjects will then be randomized in a 1:1:1 ratio to D-2570 or placebo . They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.
  Arms: placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled clinical trial. The target population is patients with moderately to severely active ulcerative colitis. A total of 120 subjects are planned to be included.

DETAILED DESCRIPTION:
The study is divided into two parts, Part A and Part B. Part A will include 30 subjects, while Part B will include 90 subjects. The primary difference between Part A and Part B is that Part A includes a single-dose pharmacokinetic (PK) study period. Other aspects, such as population selection, randomization and blinding, dosing regimens, and outcome assessments (safety and efficacy), are consistent between Part A and Part B.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria can be included in this study:

1. Subjects voluntarily take part in the study after being fully informed, sign a written informed consent form (ICF), and agree to follow procedures specified in the study protocol;
2. Males and females, 18 to 70 years of age, inclusive at the time of signing of ICF;
3. Have had an established diagnosis of ulcerative colitis (UC) of ≥ 3 months in duration prior to signing of ICF, which is supported by endoscopy reports, histopathology reports and clinical manifestations consistent with UC, as determined by investigators;
4. Involved intestinal segment extending ≥ 15 cm from the anal verge as confirmed by a screening endoscopy;
5. Active moderate to severe UC, defined by a modified Mayo score of 5 to 9 points at screening, which includes a stool frequency (SF) subscore of ≥ 2, a rectal bleeding (RB) subscore ≥ 1 and an endoscopic (ES) subscore of ≥ 2 (based on a screening endoscopy, confirmed by central reading);
6. Documentation of an inadequate response, loss of response, or intolerance (defined as interruption of drug due to an adverse reaction as evaluated by the investigator) to a treatment course of 1 or more of the following standard of care medications:
7. If a subject is using oral 5-ASAs, and/or oral glucocorticoids (≤ 20 mg/day of prednisone or equivalent dose, or ≤ 9 mg/day of budesonide or equivalent dose), and/or probiotics to treat UC, the dosage must remain stable for ≥ 2 weeks prior to the screening endoscopy and during the study period;
8. If 5-ASAs and glucocorticoids have already been discontinued, they must have been discontinued for ≥ 2 weeks prior to the screening endoscopy;

   * Exclusion Criteria

Subjects cannot be included in the study if any of the following exclusion criteria is met:

1. Diagnosed or suspected Crohn's disease, indeterminate colitis, fulminant colitis, toxic megacolon, microscopic colitis, ischemic colitis, radiation colitis, or colitis associated with diverticula;
2. History of colonic resection, subtotal or total colectomy, or surgical intervention for UC, or anticipated need for, as assessed by the investigator, surgical intervention for UC during the study, or with other gastrointestinal diseases or surgical histories that may affect the absorption of study treatment;
3. Current gastrointestinal dysplasia or past confirmed gastrointestinal dysplasia that has not been eradicated; For subjects diagnosed with UC for more than 8 years, a colonoscopy to screen for dysplasia should have been performed within 1 year prior to randomization or may be conducted during the screening colonoscopy.

   Subjects with a history of adenomatous polyps are eligible if the polyps have been completely removed (as documented in the medical records), and no residual polyps or evidence of dysplasia is found in the colonoscopy and histological examination at screening.
4. Previous history of serious herpes zoster/herpes simplex infection, including but not limited to disseminated herpes simplex/herpes zoster infection, generalized herpes zoster, herpetic encephalitis/meningitis, ocular herpes, recurrent herpes zoster, or other serious herpes zoster/herpes simplex infections assessed by the investigator, or presence of herpes zoster/herpes simplex infection at screening;
5. History of tuberculosis, active tuberculosis, latent tuberculosis, or clinical manifestations suggestive of tuberculosis infection; for subjects with latent tuberculosis infection (i.e., tested positive interferon-gamma release assay [IGRA] for Mycobacterium tuberculosis at screening) but without any symptoms, signs, laboratory findings, or imaging evidence of tuberculosis infection, re-screening is allowed after completing at least 4 weeks of standard preventive anti-tuberculosis treatment and evaluation by the investigator; subjects with indeterminate IGRA results must undergo a repeat test for confirmation, if the second test result is also indeterminate, the subject will be excluded from the study;
6. Test positive for human immunodeficiency virus (HIV) antibody, or syphilis antibody (that is the subject develops an active or latent syphilis infection), or positive for hepatitis C virus (HCV) antibody and hepatitis C virus ribonucleic acid (HCV RNA) test or a viral load greater than the upper limit of normal at the study site, or positive for hepatitis B surface antigen (HBsAg). For subjects who are HBsAg-negative but positive for hepatitis B core antibody (HBcAb), further hepatitis B virus deoxyribonucleic acid (HBV DNA) test is required. If HBV DNA is tested positive or the viral load exceeds the upper limit of normal at the study site, they will also be excluded;
7. Previous administration of a live vaccine within 3 months or an inactivated vaccine within 30 days prior to randomization, or planning to administer a live vaccine during the study or within 1 month after the last dose of investigational product;
8. Have undergone a major surgery within 8 weeks prior to randomization, or planning to undergo any surgery during the study, unless the investigator determines that the surgery will not increase the subject's risk or affect his/her ability to receive study treatment and comply with the study requirements;
9. History of a serious viral, bacterial, or fungal infection which requires intravenous (IV) anti-infectives, or hospitalization for treatment within 3 months prior to randomization, or develops a viral, bacterial, or fungal infection which requires antibiotics/anti-viral treatment within 2 weeks prior to randomization;
10. History of stool positive for C. difficile test or evidence for other enteric pathogen infections within 3 months prior to randomization or at screening. Subjects may be re-screened 30 days after completion of a standard of care course with anti-infectives, and subsequent negative testing for corresponding tests and no persistent symptoms of infection with the pathogen, upon evaluation by the investigator;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving clinical remission at Week 12 of treatment. | Week 12
  Definition of clinical remission: Based on the modified Mayo score including stool frequency subscore, rectal bleeding subscore, and endoscopic subscore. All the following criteria must be met:
  Stool frequency (SF) subscore ≤ 1, with a ≥1-point decrease from baseline; Rectal bleeding (RB) subscore = 0; Endoscopic subscore (ES) ≤ 1.

SECONDARY OUTCOMES:
Proportion of subjects achieving clinical response at Week 12 of treatment; | Week 12
● Proportion of subjects achieving symptomatic remission at 4, 8, 12 weeks of treatment; | 4, 8, 12 weeks
RB subscore change from baseline at 4, 8, 12 weeks of treatment; | 4, 8, 12 weeks
SF subscore change from baseline at 4, 8, 12 weeks of treatment; | 4, 8, 12 weeks
Proportion of subjects achieving endoscopic improvement at 12 weeks of treatment. | Week 12
Proportion of subjects achieving ES of 0 at 12 weeks of treatment; | Week 12
ES change from baseline at 12 weeks of treatment; | Week 12
Proportion of subjects with normal fecal calprotectin at 4, 8, 12 weeks of treatment; | 4, 8, 12 weeks
Proportion of subjects with normal C-reactive protein at 4, 8, 12 weeks of treatment; | 4, 8, 12 weeks
Plasma concentrations of D-2570 | 0-week 12
safety（AEs） | 0-week12
  An Adverse Event (AE) is definedas any new untoward medicaloccurrence or worsening of a preexistingmedical condition in a clinicalinvestigation participant administeredstudy treatment and that does notnecessarily have a causal relationshipwith this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: qian Cao, phD, Principal Investigator — Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine
Locations (1):
- Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No